CLINICAL TRIAL: NCT02662764
Title: A Multicenter, Open-Label Trial to Evaluate the Overall Performance of the Zalviso System™ (Sufentanil Sublingual Tablet System) 15 mcg
Brief Title: Study to Evaluate the Overall Performance of the Zalviso System™ (Sufentanil Sublingual Tablet System) 15 mcg
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Talphera, Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IAP312
Record Dates: First submitted 2016-01-20; First posted 2016-01-26 (Estimated); Results first posted 2018-08-08 (Actual); Last update posted 2018-08-08 (Actual); Status verified 2018-08

CONDITIONS: Moderate-to-severe Acute Pain
MeSH Terms: interventions — Sufentanil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes

ARMS (1):
- Zalviso™ 15 mcg (Experimental): Zalviso™(sufentanil sublingual tablet system) 15 mcg
  Interventions: Drug: Zalviso™ 15 mcg

INTERVENTIONS:
Drug: Zalviso™ 15 mcg — Zalviso™ (sufentanil sublingual tablet system) 15 mcg. Tablets to be self-administered by the patient as needed for pain, no more than every 20 minutes, for 24 hours and up to 72 hours
  Other Names: Zalviso™ (sufentanil sublingual tablet system) 15 mcg

SUMMARY:
Study to evaluate the overall performance of the Zalviso System™ (sufentanil sublingual tablet system) 15 mcg

DETAILED DESCRIPTION:
320 adult postoperative in-patients, who met all study entry requirements, and were expected to require opioid analgesia for at least 24 hours, and up to 72 hours, after surgery were enrolled. Patients used the Zalviso™ (sufentanil sublingual tablet system) 15 mcg to self-administer a tablet of study drug as needed for pain. The System was evaluated for usability and functionality for up to 72 hours.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients who were 18 years of age or older.
2. Patients who were scheduled to undergo surgery under general or spinal anesthesia that does not include intrathecal opioids during the operation.
3. Patients classified as American Society of Anesthesiologists (ASA) class I - III (Appendix I).
4. Female patients of childbearing potential must have been using an effective method of birth control at the time of screening visit and for 30 days following the end of the study period. Acceptable methods of birth control included oral or transdermal contraceptives, condom, spermicidal foam, intrauterine device (IUD), progestin implant or injection, abstinence, vaginal ring, or sterilization of partner. The reason for non-child bearing potential, such as bilateral tubal ligation, bilateral oophorectomy, hysterectomy, or postmenopausal for > 1 year, was specified. Patients using hormonal forms of contraception were also willing to use a barrier method of contraception from screening through 30 days following the study period.
5. Post-surgical patients who had been admitted to the PACU, and were expected to have acute pain requiring opioids for 24 - 72 hours after surgery.

Exclusion Criteria:

1. Patients who had taken an opioid for more than 30 consecutive days, at a daily dose of 15 mg or more of morphine (or equivalent), within the past 3 months prior to surgery (e.g. more than 3 doses per day of Vicodin®, Norco®, Lortab® with 5 mg hydrocodone per tablet).
2. Patients who were currently taking monoamine oxidase inhibitors (MAOIs) or had taken MAOIs within 14 days of the first dose of study drug.
3. Patients with current sleep apnea that had been documented by a sleep laboratory study or were on home continuous positive airway pressure (CPAP).
4. Patients with an allergy or hypersensitivity to opioids.
5. Patients who were currently taking monoamine oxidase inhibitors (MAOIs) or had taken MAOIs within 14 days of the first dose of study drug.
6. Patients with current sleep apnea that had been documented by a sleep laboratory study or were on home continuous positive airway pressure (CPAP).
7. Patients who were receiving oxygen therapy at the time of screening.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 320 (Actual)
Dates: Start 2016-09-28 (Actual); Primary Completion 2017-04-14 (Actual); Study Completion 2017-05-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pamela Palmer, MD, PhD, Study Director — Talphera, Inc
Locations (11):
- United States (11):
  - Eliza Coffee Memorial Hospital, Florence, Alabama
  - Shoals Medical Trials, Sheffield, Alabama
  - Arizona Research Center, Phoenix, Arizona
  - Gulfcoast Research Associates, Sarasota, Florida
  - G&G Research, Vero Beach, Florida
  - Orthopedic Center of Vero Beach, Vero Beach, Florida
  - Visions Clinical Research, Wellington, Florida
  - Southeastern Center for Clinical Trials, Decatur, Georgia
  - Westside Surgical Hospital, Houston, Texas
  - Hermann Drive Surgical Hospital, Houston, Texas
  - Jean Brown Research, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Zalviso™ 15 mcg
Started | 320
Completed | 290 (First 24-hours of study treatment)
Not Completed | 30
Not completed — Adverse Event | 6
Not completed — Lack of Efficacy | 8
Not completed — Protocol Violation | 1
Not completed — Withdrawal by Subject | 5
Not completed — Device failure | 4
Not completed — Patient changed treatment | 1
Not completed — Patient discharged prior to 24 hrs | 5

BASELINE CHARACTERISTICS:
Arm/Group | Zalviso™ 15 mcg
Number analyzed (Participants) | 320
Age, Customized [Count of Participants; unit: Participants]
  Age, Customized: <65 | 198
  Age, Customized: > or equal to 65 | 122
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 193
  Male | 127
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 18
  Not Hispanic or Latino | 302
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 35
  White | 280
  More than one race | 1
  Unknown or Not Reported | 1

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients Who Experienced at Least One System-generated Error Based on the Controller Data While Using the Zalviso System
Time Frame: Up to 72 hours
Measure: Number; unit: percentage of patients
Arm/Group | Zalviso™ 15 mcg
Number analyzed (Participants) | 320
percentage of patients | 2.2

2. Primary Outcome: Percentage of Patients, if Any, With Tablets Dispensed But Not Requested
Time Frame: Up to 72 hours
Measure: Number; unit: percentage of patients
Groups:
- Zalviso™ 15 mcg: Zalviso™(sufentanil sublingual tablet system) 15 mcg
  Zalviso™ 15 mcg: Zalviso™ (sufentanil sublingual tablet system) 15 mcg. Tablets to be self-administered by the patient as needed for pain, no more than every 20 minutes, for up to 72 hours
Arm/Group | Zalviso™ 15 mcg
Number analyzed (Participants) | 320
percentage of patients | 0

3. Primary Outcome: Percentage of Patients, if Any, With Tablet Dispensed When the Zalviso System Was in Lockout
Time Frame: Up to 72 hours
Measure: Number; unit: percentage of patients
Arm/Group | Zalviso™ 15 mcg
Number analyzed (Participants) | 320
percentage of patients | 0

4. Primary Outcome: Percentage of Patients With Misplaced Tablet(s)
Time Frame: Up to 72 hours
Measure: Number; unit: percentage of patients
Arm/Group | Zalviso™ 15 mcg
Number analyzed (Participants) | 320
percentage of patients | 3.8

5. Primary Outcome: Number of Misplaced Tablets (i.e., Tablet Found Outside the Patient's Mouth)
Time Frame: Up to 24 hours
Measure: Number; unit: tablets
Groups:
- Zalviso™ 15 mcg: Zalviso™ 15 mcg: Zalviso™ (sufentanil sublingual tablet system) 15 mcg. Tablets to be self-administered by the patient as needed for pain, no more than every 20 minutes, for 24 hours.
Arm/Group | Zalviso™ 15 mcg
Number analyzed (Participants) | 320
tablets | 13

6. Primary Outcome: Percentage of Patients Who Experienced Either a System-generated Error or a Misplaced Tablet (i.e., a Dispense Failure)
Time Frame: Up to 72 hours
Measure: Number; unit: percentage of patients
Arm/Group | Zalviso™ 15 mcg
Number analyzed (Participants) | 320
percentage of patients | 5.6

7. Primary Outcome: Number of Zalviso System Notifications to the Nurse to Retrain Patient to Not Pull Down on the Controller While Dosing
Time Frame: Up to 72 hours
Measure: Number; unit: Notifications
Arm/Group | Zalviso™ 15 mcg
Number analyzed (Participants) | 320
Notifications | 0

8. Primary Outcome: Percentage of Patients Who Experienced at Least One System-generated Error Based on the Controller Data While Using the Zalviso System
Time Frame: Up to 72 hours
Measure: Number; unit: percentage of patients
Arm/Group | Zalviso™ 15 mcg
Number analyzed (Participants) | 320
percentage of patients | 2.2

9. Primary Outcome: Percentage of Patients Who Experienced Either a System-generated Error or a Misplaced Tablet That Caused an Analgesic Gap
Time Frame: Up to 72 hours
Measure: Number; unit: percentage of participants
Arm/Group | Zalviso™ 15 mcg
Number analyzed (Participants) | 320
percentage of participants | 2.8

10. Primary Outcome: Percentage of Patients Who Rate the Patient Global Assessment (PGA) of Method of Pain Control Over 24 Hours as "Good" or "Excellent"
Time Frame: Up to 24 hours
Population: This assessment was completed by patients who were not sleeping at the time of the assessment, had not withdrawn prematurely, or for whom the assessment was not done in error.
Measure: Number; unit: percentage of patients
Arm/Group | Zalviso™ 15 mcg
Number analyzed (Participants) | 320
percentage of patients | 86.1

11. Primary Outcome: Percentage of Patients Who Rate the Patient Global Assessment (PGA) of Method of Pain Control Over 48 Hours as "Good" or "Excellent"
Time Frame: Up to 48 hours
Population: This assessment completed by patients who were not sleeping at the time of the assessment, had not withdrawn prematurely, or for whom the assessment was not done in error.
Measure: Number; unit: percentage of patients
Arm/Group | Zalviso™ 15 mcg
Number analyzed (Participants) | 113
percentage of patients | 88.5

12. Primary Outcome: Percentage of Patients Who Rate the Patient Global Assessment (PGA) of Method of Pain Control Over 72 Hours as "Good" or "Excellent"
Time Frame: Up to 72 hours
Population: as for outcome 10
Measure: Number; unit: percentage of patients
Arm/Group | Zalviso™ 15 mcg
Number analyzed (Participants) | 14
percentage of patients | 100

13. Primary Outcome: Percentage of Patients Who Responded to the Patient Global Assessment (PGA) as "Poor" at 24 Hours
Time Frame: Up to 24 hours
Population: This assessment was completed by subjects who were not sleeping at the time of the assessment, had not withdrawn prematurely, or for whom the assessment was not done in error.
Measure: Number; unit: percentage of patients
Arm/Group | Zalviso™ 15 mcg
Number analyzed (Participants) | 294
percentage of patients | 1.4

14. Primary Outcome: Percentage of Patients Who Responded to the Patient Global Assessment (PGA) as "Fair" at 24 Hours
Time Frame: Up to 24 hours
Population: as for outcome 10
Measure: Number; unit: percentage of patients
Arm/Group | Zalviso™ 15 mcg
Number analyzed (Participants) | 294
percentage of patients | 12.6

15. Primary Outcome: Percentage of Patients Who Responded to the Patient Global Assessment (PGA) as "Good" at 24 Hours
Time Frame: Up to 24 hours
Population: as for outcome 10
Measure: Number; unit: percentage of patients
Arm/Group | Zalviso™ 15 mcg
Number analyzed (Participants) | 294
percentage of patients | 40.8

16. Primary Outcome: Percentage of Patients Who Responded to the Patient Global Assessment (PGA) as "Excellent" at 24 Hours
Time Frame: Up to 24 hours
Population: as for outcome 10
Measure: Number; unit: percentage of patients
Arm/Group | Zalviso™ 15 mcg
Number analyzed (Participants) | 294
percentage of patients | 45.2

17. Primary Outcome: Percentage of Patients Who Responded to the Patient Global Assessment (PGA) at 48 Hours as "Poor"
Time Frame: Up to 48 hours
Population: as for outcome 13
Measure: Number; unit: percentage of patients
Arm/Group | Zalviso™ 15 mcg
Number analyzed (Participants) | 113
percentage of patients | 0.9

18. Primary Outcome: Percentage of Patients Who Responded to the Patient Global Assessment (PGA) at 48 Hours as "Fair"
Time Frame: Up to 48 hours
Population: as for outcome 10
Measure: Number; unit: percentage of patients
Arm/Group | Zalviso™ 15 mcg
Number analyzed (Participants) | 113
percentage of patients | 10.6

19. Primary Outcome: Percentage of Patients Who Responded to the Patient Global Assessment (PGA) at 48 Hours as "Good"
Time Frame: Up to 48 hours
Population: as for outcome 10
Measure: Number; unit: percentage of patients
Arm/Group | Zalviso™ 15 mcg
Number analyzed (Participants) | 113
percentage of patients | 41.6

20. Primary Outcome: Percentage of Patients Who Responded to the Patient Global Assessment (PGA) at 48 Hours as "Excellent"
Time Frame: Up to 48 hours
Population: as for outcome 10
Measure: Number; unit: percentage of patients
Arm/Group | Zalviso™ 15 mcg
Number analyzed (Participants) | 113
percentage of patients | 46.9

21. Primary Outcome: Percentage of Patients Who Responded to the Patient Global Assessment (PGA) at 72 Hours as "Poor"
Time Frame: Up to 72 hours
Population: as for outcome 10
Measure: Number; unit: percentage of patients
Arm/Group | Zalviso™ 15 mcg
Number analyzed (Participants) | 14
percentage of patients | 0

22. Primary Outcome: Percentage of Patients Who Responded to the Patient Global Assessment (PGA) at 72 Hours as "Fair"
Time Frame: Up to 72 hours
Population: as for outcome 10
Measure: Number; unit: percentage of patients
Arm/Group | Zalviso™ 15 mcg
Number analyzed (Participants) | 14
percentage of patients | 0

23. Primary Outcome: Percentage of Patients Who Responded to the Patient Global Assessment (PGA) at 72 Hours as "Good"
Time Frame: Up to 72 hours
Population: as for outcome 13
Measure: Number; unit: percentage of patients
Arm/Group | Zalviso™ 15 mcg
Number analyzed (Participants) | 14
percentage of patients | 42.9

24. Primary Outcome: Percentage of Patients Who Responded to the Patient Global Assessment (PGA) at 72 Hours as "Excellent"
Time Frame: Up to 72 hours
Population: as for outcome 10
Measure: Number; unit: percentage of patients
Arm/Group | Zalviso™ 15 mcg
Number analyzed (Participants) | 14
percentage of patients | 57.1

25. Primary Outcome: Percentage of Healthcare Professionals (HCPs) Who Rated the Healthcare Professional Global Assessment (HPGA) of Method of Pain Control Over 24 Hours as "Good" or "Excellent"
Time Frame: Up to 24 hours
Population: Overall number of HCPs who completed the assessment. On rare occasions, the HCP did not complete the assessment in error.
Measure: Number; unit: percentage of HCPs
Arm/Group | Zalviso™ 15 mcg
Number analyzed (Participants) | 270
percentage of HCPs | 91.1

26. Primary Outcome: Percentage of Healthcare Professionals (HCPs) Who Rate the Healthcare Professional Global Assessment (HPGA) of Method of Pain Control Over 48 Hours as "Good" or "Excellent"
Time Frame: Up to 48 hours
Population: as for outcome 25
Measure: Number; unit: percentage of HCPs
Arm/Group | Zalviso™ 15 mcg
Number analyzed (Participants) | 102
percentage of HCPs | 95.1

27. Primary Outcome: Percentage of Healthcare Professionals (HCPs) Who Rated the Healthcare Professional Global Assessment (HPGA) of Method of Pain Control Over 72 Hours as "Good" or "Excellent"
Time Frame: Up to 72 hours
Population: Overall number of HCPs who completed the assessment. In rare cases, the HCP did not complete the assessment in error.
Measure: Number; unit: percentage of HCPs
Arm/Group | Zalviso™ 15 mcg
Number analyzed (Participants) | 12
percentage of HCPs | 100

28. Primary Outcome: Percentage of Healthcare Professional (HCPs) Who Responded to the Healthcare Professional Global Assessment (HPGA) as "Poor" at 24 Hours
Time Frame: Up to 24 hours
Population: as for outcome 25
Measure: Number; unit: percentage of HCPs
Arm/Group | Zalviso™ 15 mcg
Number analyzed (Participants) | 270
percentage of HCPs | 0.7

29. Primary Outcome: Percentage of Healthcare Professional Global Assessment (HCPs) Who Responded to the Healthcare Professional Global Assessment (HPGA) as "Fair" at 24 Hours
Time Frame: Up to 24 hours
Population: as for outcome 25
Measure: Number; unit: percentage of HCPs
Arm/Group | Zalviso™ 15 mcg
Number analyzed (Participants) | 270
percentage of HCPs | 8.1

30. Primary Outcome: Percentage of Healthcare Professionals (HCPs) Who Responded to the Healthcare Professional Global Assessment (HPGA) as "Good" at 24 Hours
Time Frame: Up to 24 hours
Population: as for outcome 25
Measure: Number; unit: percentage of HCPs
Arm/Group | Zalviso™ 15 mcg
Number analyzed (Participants) | 270
percentage of HCPs | 38.9

31. Primary Outcome: Percentage of Healthcare Professional (HCPs) Who Responded to the Healthcare Professional Global Assessment (HPGA) as "Excellent" at 24 Hours
Time Frame: Up to 24 hours
Population: as for outcome 25
Measure: Number; unit: percentage of HCPs
Arm/Group | Zalviso™ 15 mcg
Number analyzed (Participants) | 270
percentage of HCPs | 52.2

32. Primary Outcome: Percentage of Healthcare Professionals (HCPs) Who Responded to the Healthcare Professional Global Assessment (HPGA) at 48 Hours as "Poor"
Time Frame: Up to 48 hours
Population: as for outcome 25
Measure: Number; unit: percentage of HCPs
Arm/Group | Zalviso™ 15 mcg
Number analyzed (Participants) | 102
percentage of HCPs | 1.0

33. Primary Outcome: Percentage of Healthcare Professionals (HCPs) Who Responded to the Healthcare Professional Global Assessment (HPGA) at 48 Hours as "Fair"
Time Frame: Up to 48 hours
Population: as for outcome 25
Measure: Number; unit: percentage of HCPs
Arm/Group | Zalviso™ 15 mcg
Number analyzed (Participants) | 102
percentage of HCPs | 3.9

34. Primary Outcome: Percentage of Healthcare Professionals (HCPs) Who Responded to the Healthcare Professional Global Assessment (HPGA )at 48 Hours as "Good"
Time Frame: Up to 48 hours
Population: as for outcome 25
Measure: Number; unit: percentage of HCPs
Arm/Group | Zalviso™ 15 mcg
Number analyzed (Participants) | 102
percentage of HCPs | 27.5

35. Primary Outcome: Percentage of Healthcare Professionals (HCPs) Who Responded to the Healthcare Professional Global Assessment (HPGA) at 48 Hours as "Excellent"
Time Frame: Up to 48 hours
Population: as for outcome 25
Measure: Number; unit: percentage of HCPs
Arm/Group | Zalviso™ 15 mcg
Number analyzed (Participants) | 102
percentage of HCPs | 67.6

36. Primary Outcome: Percentage of Healthcare Professionals (HCPs) Who Responded to the Healthcare Professional Global Assessment (HPGA) at 72 Hours as "Poor"
Time Frame: Up to 72 hours
Population: as for outcome 25
Measure: Number; unit: percentage of HCPs
Arm/Group | Zalviso™ 15 mcg
Number analyzed (Participants) | 12
percentage of HCPs | 0

37. Primary Outcome: Percentage of Healthcare Professionals (HCPs) Who Responded to the Healthcare Professional Global Assessment (HPGA) at 72 Hours as "Fair"
Time Frame: Up to 72 hours
Population: as for outcome 25
Measure: Number; unit: percentage of HCPs
Groups:
- Zalviso™ 15 mcg: Zalviso™ 15 mcg: Zalviso™ (sufentanil sublingual tablet system) 15 mcg. Tablets to be self-administered by the patient as needed for pain, no more than every 20 minutes, for at least 24 hours and up to 72 hours.
Arm/Group | Zalviso™ 15 mcg
Number analyzed (Participants) | 12
percentage of HCPs | 0

38. Primary Outcome: Percentage of Healthcare Professionals (HCPs) Who Responded to the Healthcare Professional Global Assessment (HPGA) at 72 Hours as "Good"
Time Frame: Up to 72 hours
Population: as for outcome 25
Measure: Number; unit: percentage of HCPs
Arm/Group | Zalviso™ 15 mcg
Number analyzed (Participants) | 12
percentage of HCPs | 8.3

39. Primary Outcome: Percentage of Healthcare Professionals (HCPs) Who Responded to the Healthcare Professional Global Assessment (HPGA) at 72 Hours as "Excellent"
Time Frame: Up to 72 hours
Population: as for outcome 25
Measure: Number; unit: percentage of HCPs
Arm/Group | Zalviso™ 15 mcg
Number analyzed (Participants) | 12
percentage of HCPs | 91.7

40. Primary Outcome: Percentage of Patients Who Terminated From the Study Due to Inadequate Analgesia Over the 24-hour Study Period
Time Frame: Up to 24 hours
Measure: Number; unit: percentage of patients
Arm/Group | Zalviso™ 15 mcg
Number analyzed (Participants) | 320
percentage of patients | 2.5

41. Primary Outcome: Percentage of Patients Who Terminated From the Study Due to Inadequate Analgesia After the 24-hour Study Period and Prior to or During the 48 Hour Study Period
Time Frame: Up to 48 hours
Measure: Number; unit: percentage of patients
Arm/Group | Zalviso™ 15 mcg
Number analyzed (Participants) | 290
percentage of patients | 2.8

42. Primary Outcome: Percentage of Patients Who Terminated From the Study Due to Inadequate Analgesia Prior to or During the 72 Hour Study Period
Time Frame: Up to 72 hours
Measure: Number; unit: percentage of patients
Arm/Group | Zalviso™ 15 mcg
Number analyzed (Participants) | 93
percentage of patients | 0

43. Primary Outcome: Time-weighted Summed Pain Intensity Difference (SPID) Over the 24-hour Study Period (SPID24)
Description: The pain intensity difference (PID) at each evaluation time point after the dose of study drug is the difference in pain intensity at the specific evaluation time point and baseline pain intensity [PID(evaluation time after the first dose) = PI(baseline) - PI(evaluation time after the first dose)]. A pain intensity score ranging from 0 (no pain) to 10 (worst possible pain) is obtained at baseline and at protocol-specified time points throughout the 24 hour period. The time-weighted SPID24 is the time-weighted summed PID over the 24-hour study period. A negative score indicates an increase in pain intensity and a higher score indicates a greater decrease in pain intensity.The scores ranged from - 72 to 204.
Time Frame: Up to 24 hours
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Zalviso™ 15 mcg
Number analyzed (Participants) | 313
units on a scale | 63.09 (2.58)

44. Primary Outcome: Time-weighted Summed Pain Intensity Difference (SPID) Over the 48-hour Study Period (SPID-48) Study Period
Description: The pain intensity difference (PID) at each evaluation time point after the dose of study drug is the difference in pain intensity at the specific evaluation time point and baseline pain intensity [PID(evaluation time after the first dose) = PI(baseline) - PI(evaluation time after the first dose)]. A pain intensity score ranging from 0 (no pain) to 10 (worst possible pain) is obtained at baseline and at protocol-specified time points and throughout the 48 hour period. The time-weighted SPID48 is the time-weighted summed PID over the 48-hour study period. A negative score indicates an increase in pain intensity and a higher score indicates a greater decrease in pain intensity.The scores ranged from -144 to 408.
Time Frame: Up to 48 hours
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Zalviso™ 15 mcg
Number analyzed (Participants) | 313
units on a scale | 130.69 (5.56)

45. Primary Outcome: Time-weighted Summed Pain Intensity Difference (SPID) Over the 72-hour Study Period (SPID-72) Study Period
Description: The pain intensity difference (PID) at each evaluation time point after the dose of study drug is the difference in pain intensity at the specific evaluation time point and baseline pain intensity [PID(evaluation time after the first dose) = PI(baseline) - PI(evaluation time after the first dose)]. A pain intensity score ranging from 0 (no pain) to 10 (worst possible pain) is obtained at baseline and at protocol-specified time points throughout the 72 hour period. The time-weighted SPID72 is the time-weighted summed PID over the 72-hour study period. A negative score indicates an increase in pain intensity and a higher score indicates a greater decrease in pain intensity. The scores ranged from -239 to 624.
Time Frame: Up to 72 hours
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Zalviso™ 15 mcg
Number analyzed (Participants) | 313
units on a scale | 204.66 (8.61)

46. Primary Outcome: Total Pain Relief (TOTPAR) Over the 24-hour Study Period (TOTPAR24)
Description: Total pain relief over the 24-hour study period. A higher TOTPAR score means a greater relief in pain. Range of scores was from 0.00 to 96.00.
Time Frame: Up to 24 hours
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Zalviso™ 15 mcg
Number analyzed (Participants) | 318
units on a scale | 54.27 (1.14)

47. Primary Outcome: Total Pain Relief (TOTPAR) Over the 48-hour Study Period (TOTPAR48)
Description: Total pain relief over the 48-hour study period. A higher TOTPAR score means a greater relief in pain. Range of scores was from 0.00 to 192.00.
Time Frame: Up to 48 hours
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Zalviso™ 15 mcg
Number analyzed (Participants) | 318
units on a scale | 111.42 (2.35)

48. Primary Outcome: Total Pain Relief (TOTPAR) Over the 72-hour Study Period (TOTPAR72)
Description: Total pain relief over the 72-hour study period. A higher TOTPAR means a greater relief in pain. Range of scores was from 0.00 to 288.00.
Time Frame: Up to 72 hours
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Zalviso™ 15 mcg
Number analyzed (Participants) | 318
units on a scale | 171.10 (3.70)

49. Primary Outcome: Pain Intensity (PI) at Each Evaluation Time Point
Description: At protocol-specified time points, the patient is asked to self-record his/her current level of pain on an 11-point numerical rating scale where 0 equals no pain and 10 equals the worst possible pain.
Time Frame: Up to 72 hours
Population: as for outcome 10
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Zalviso™ 15 mcg
Number analyzed (Participants) | 313
units on a scale
  Baseline | 5.84 (0.07)
  15 minutes | 4.77 (0.13)
  30 minutes | 4.46 (0.13)
  45 minutes | 4.05 (0.13)
  1 hour | 3.70 (0.13)
  2 hours | 3.37 (0.12)
  4 hours | 3.39 (0.12)
  6 hours | 3.20 (0.12)
  8 hours | 3.18 (0.13)
  10 hours | 3.10 (0.13)
  12 hours | 2.97 (0.12)
  16 hours | 3.08 (0.13)
  20 hours | 3.20 (0.14)
  24 hours | 3.16 (0.13)
  28 hours | 3.16 (0.13)
  32 hours | 3.15 (0.13)
  36 hours | 3.06 (0.13)
  40 hours | 2.96 (0.13)
  44 hours | 2.93 (0.13)
  48 hours | 2.82 (0.13)
  52 hours | 2.76 (0.12)
  56 hours | 2.77 (0.12)
  60 hours | 2.75 (0.12)
  64 hours | 2.76 (0.12)
  68 hours | 2.77 (0.12)
  72 hours | 2.76 (0.12)

50. Primary Outcome: Pain Intensity Difference (PID) at Each Evaluation Time Point
Description: The PID at each evaluation time point after the dose of study drug is the difference in pain intensity at the specific evaluation time point and baseline pain intensity [PID(evaluation time after the first dose) = PI(baseline) - PI(evaluation time after the first dose)]. The higher the PID score, the lower the pain intensity. The scores ranged from - 239 to 624.
Time Frame: Up to 72 hours
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Zalviso™ 15 mcg
Number analyzed (Participants) | 313
units on a scale
  Baseline | 5.84 (0.07)
  15 minutes | 1.07 (0.10)
  30 minutes | 1.38 (0.10)
  45 minutes | 1.79 (0.11)
  1 hour | 2.14 (0.11)
  2 hours | 2.48 (0.12)
  4 hours | 2.45 (0.13)
  6 hours | 2.64 (0.12)
  8 hours | 2.67 (0.13)
  10 hours | 2.74 (0.13)
  12 hours | 2.88 (0.12)
  16 hours | 2.77 (0.13)
  20 hours | 2.65 (0.14)
  24 hours | 2.69 (0.14)
  28 hours | 2.68 (0.14)
  32 hours | 2.69 (0.14)
  36 hours | 2.78 (0.14)
  40 hours | 2.88 (0.14)
  44 hours | 2.91 (0.14)
  48 hours | 3.02 (0.14)
  52 hours | 3.08 (0.14)
  56 hours | 3.08 (0.13)
  60 hours | 3.09 (0.14)
  64 hours | 3.08 (0.13)
  68 hours | 3.08 (0.13)
  72 hours | 3.08 (0.13)

51. Primary Outcome: Pain Relief (PR) at Each Evaluation Time Point
Description: At protocol-specified time points, the patient is asked to self-record his/her current level of pain relief on 5-point numerical rating scale where 0 equaled no pain relief and 4 equaled complete pain relief. The baseline score references the baseline pain intensity score and the following timepoints reference pain relief scores.
Time Frame: Up to 72 hours
Population: as for outcome 10
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Zalviso™ 15 mcg
Number analyzed (Participants) | 318
units on a scale
  (Not Applicable): number analyzed (Participants) | 312
  (Not Applicable) | NA (NA) — Pain relief was not collected at baseline since the patient had not yet received study drug
  15 minutes: number analyzed (Participants) | 310
  15 minutes | 1.18 (0.07)
  30 minutes: number analyzed (Participants) | 317
  30 minutes | 1.42 (0.06)
  45 minutes: number analyzed (Participants) | 317
  45 minutes | 1.67 (0.06)
  1 hour: number analyzed (Participants) | 317
  1 hour | 1.81 (0.07)
  2 hours | 2.08 (0.06)
  4 hours | 2.12 (0.06)
  6 hours | 2.24 (0.06)
  8 hours | 2.24 (0.06)
  10 hours | 2.32 (0.06)
  12 hours | 2.37 (0.06)
  16 hours | 2.31 (0.06)
  20 hours | 2.30 (0.06)
  24 hours | 2.42 (0.06)
  28 hours | 2.37 (0.06)
  32 hours | 2.34 (0.06)
  36 hours | 2.34 (0.06)
  40 hours | 2.39 (0.06)
  44 hours | 2.41 (0.06)
  48 hours | 2.44 (0.06)
  52 hours | 2.48 (0.06)
  56 hours | 2.48 (0.06)
  60 hours | 2.49 (0.06)
  64 hours | 2.48 (0.06)
  68 hours | 2.49 (0.06)
  72 hours | 2.50 (0.06)

52. Primary Outcome: Patient Usability Questionnaire (PUQ)
Description: Questionnaire completed by patients at the end of his/her participation in the study regarding the usability of Zalviso.
Time Frame: Up to 72 hours
Measure: Number; unit: percentage of patients
Arm/Group | Zalviso™ 15 mcg
Number analyzed (Participants) | 317
percentage of patients
  Agreed Zalviso was easy to use | 90.5
  Agreed having confidence to dose | 92.4
  Agreed Zalviso worked consistently as expected | 82.3
  Agreed they knew how to use Zalviso | 93.4
  Agreed they knew what to do if a tablet dropped | 86.1
  Agreed Zalviso instructions were explained | 91.2
  Agreed to request Zalviso after next surgery | 80.4

53. Primary Outcome: Nurse Usability Questionnaire (NUQ)
Description: Questionnaire regarding the usability of Zalviso completed by HCPs who had set up at least 5 Zalviso Systems for patients
Time Frame: Up to 72 hours
Measure: Number; unit: percentage of HCPs
Arm/Group | Zalviso™ 15 mcg
Number analyzed (Participants) | 40
percentage of HCPs
  Agreed Zalviso easy to set up | 92.5
  Agreed had confidence to set up Zalviso | 92.5
  Agreed no need to trouble-shoot during patient use | 87.5
  Agreed with appropriate tablet accountability | 100
  Agreed Zalviso was not time-consuming to set up | 72.5
  Agreed Zalviso instructions were clear | 90
  Would recommend using Zalviso | 87.5

54. Primary Outcome: Number of Study Drug Doses Used
Time Frame: Up to 72 hours
Measure: Mean (Standard Deviation); unit: doses
Arm/Group | Zalviso™ 15 mcg
Number analyzed (Participants) | 320
doses
  24-hour treatment period | 15.7 (9.9)
  48-hour treatment period | 21.9 (14.8)
  72-hour treatment period | 22.8 (15.7)

55. Primary Outcome: Average Hourly Use of Study Drug
Description: Average number of study drug doses used per hour, adjusting by treatment exposure time and study period
Time Frame: Up to 72 hours
Measure: Mean (Standard Deviation); unit: average number of study doses per hour
Arm/Group | Zalviso™ 15 mcg
Number analyzed (Participants) | 320
average number of study doses per hour | 0.82 (0.51)

56. Primary Outcome: Average Inter-dosing Interval (in Minutes)
Time Frame: Up to 72 hours
Measure: Mean (Standard Deviation); unit: average interval (minutes) between doses
Arm/Group | Zalviso™ 15 mcg
Number analyzed (Participants) | 316
average interval (minutes) between doses
  24-hour study period | 121.4 (116.2)
  48-hour study period | 123.2 (151.6)
  72-hour study period | 120.9 (109.7)

57. Primary Outcome: Total Amount of Supplemental Morphine (mg) Utilized
Description: Supplemental opioid medication (2 mg IV morphine) was allowed in the first 30 minutes after the first on-demand dose of study drug had been administered, if necessary, to keep a patient comfortable. Otherwise, supplemental opioid medication (2 mg IV morphine, no more frequently than hourly) was allowed for pain due to ambulation or with the initiation of passive range of motion therapy throughout the remainder of the study.
Time Frame: Up to 72 hours
Population: Amount of supplemental morphine (mg) utilized by patients
Measure: Mean (Standard Deviation); unit: amount of morphine (mg) used
Arm/Group | Zalviso™ 15 mcg
Number analyzed (Participants) | 320
amount of morphine (mg) used | 0.1 (0.4)

ADVERSE EVENTS:
Time Frame: From the time of first study medication dose through 72 hours, including those reported 12 hours after the last dose was taken
Arm/Group | Zalviso™ 15 mcg
All-Cause Mortality (participants affected / at risk) | 0/320
Serious Adverse Events (participants affected / at risk) | 3/320
Other Adverse Events (participants affected / at risk) | 190/320
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Zalviso™ 15 mcg (N=320)
Anaemia (Blood and lymphatic system disorders) | 1 (1)
Cardiac Failure Chronic (Cardiac disorders) | 1 (1)
Pyrexia (General disorders) | 1 (1)
Renal Injury (Injury, poisoning and procedural complications) | 1 (1)
Sedation (Nervous system disorders) | 1 (1)
Hypotension (Vascular disorders) | 1 (1)
Labile blood pressure (Vascular disorders) | 1 (1)
Chronic renal failure (Renal and urinary disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Zalviso™ 15 mcg (N=320)
Bradycardia (Cardiac disorders) | 17 (34)
Tachycardia (Cardiac disorders) | 8 (8)
Nausea (Gastrointestinal disorders) | 84 (88)
Vomiting (Gastrointestinal disorders) | 32 (49)
Constipation (Gastrointestinal disorders) | 8 (8)
Oxygen saturation decreased (Investigations) | 19 (25)
Hypokalaemia (Metabolism and nutrition disorders) | 14 (14)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 25 (25)
Dizziness (Nervous system disorders) | 14 (16)
Headache (Nervous system disorders) | 12 (13)
Pruritis (Skin and subcutaneous tissue disorders) | 11 (11)
Hypotension (Vascular disorders) | 36 (113)
Pyrexia (General disorders) | 10 (10)
Hypertension (Vascular disorders) | 7 (7)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Investigator must obtain approval from AcelRx in order to discuss or publish trial results

DOCUMENTS (3):
  • Statistical Analysis Plan (2017-06-10): https://cdn.clinicaltrials.gov/large-docs/64/NCT02662764/SAP_000.pdf
  • Informed Consent Form (2016-01-19): https://cdn.clinicaltrials.gov/large-docs/64/NCT02662764/ICF_001.pdf
  • Study Protocol (2016-01-13): https://cdn.clinicaltrials.gov/large-docs/64/NCT02662764/Prot_002.pdf